CLINICAL TRIAL: NCT07358234
Title: Prospective Trial Comparing Swallowed Topical Budesonide With Subcutaneous Dupilumab on Esophageal Diameter and Fibrotic Change in Eosinophilic Esophagitis
Brief Title: Comparison of Eohilia With Dupixent on Esophagus Diameter in Patients With Eosinophilic Esophagitis.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Diana L. Snyder, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-005776
Record Dates: First submitted 2025-12-23; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: dupilumab; budesonide oral suspension; Eohilia; Dupixent
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- budesonide oral suspension (Eohilia) (Active Comparator): 2mg twice daily
  Interventions: Drug: budesonide oral suspension
- dupilumab (Dupixent) (Active Comparator): 300 mg weekly injection
  Interventions: Drug: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT]

INTERVENTIONS:
Drug: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT] — 300 mg weekly injection
  Arms: dupilumab (Dupixent)
Drug: budesonide oral suspension — 2mg twice daily
  Other Names: Eohilia
  Arms: budesonide oral suspension (Eohilia)

SUMMARY:
The purpose of this study is to compare Eosinophilic Esophagitis treatments Eohilia with Dupixent in their effects on diameter and scarring of the esophagus.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a chronic disease mediated by environmental allergens and type 2 immune inflammation which causes significant symptoms, food impactions, and stenosis. EoE is associated with significant esophageal stricturing disease. In particular, the odds of developing fibrostenotic disease in EoE more than double per decade of life, and the longer symptoms are present prior to diagnosis and treatment, the higher the likelihood of esophageal strictures being present.

Dupilumab and budesonide oral suspension are key treatments for EoE. Dupilumab was FDA approved for EoE in 2022 and inhibits IL-4 and IL-13 signaling which mediate type-2 inflammation and may have an anti-fibrotic effect. IL-13 promotes M2 macrophage polarization, and a recent study showed fibrosis was macrophage-dependent in a mouse model of EoE. Swallowed topical steroids have been used off label in patients with EoE for several years with studies showing effects on improvement in esophageal diameter and reduction in esophageal strictures. The budesonide oral suspension was recently FDA approved in 2024. Further study is needed to understand the effect of these treatments on esophageal stenosis and fibrosis as no clinical trials have compared these treatments or their effects on esophageal diameter to date. Barium esophagram and functional lumen imaging probe (FLIP) are important tools used to measure esophageal diameter in EoE. The investigators hypothesize that dupilumab is superior to topical budesonide oral suspension for its effect on esophagram minimum diameter and FLIP distensibility plateau in EoE patients.

• Primary Efficacy Endpoint:

Alternative Hypothesis: There will be a greater increase in minimum esophageal diameter in patients receiving dupilumab compared to budesonide oral suspension at 12 weeks.

• Secondary Efficacy Endpoint(s):

Alternative Hypothesis: There will be greater distensibility on EndoFLIP topography in patients receiving dupilumab compared to budesonide oral suspension at 12 weeks. Symptoms, endoscopic findings, and histologic severity will be improved in patients receiving dupilumab compared to budesonide oral suspension at 12 weeks. Lamina propria fibrosis and collagen fiber density as determined by second harmonic generation microscopy will be improved in the dupilumab group in comparison to the budesonide oral suspension group.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged ≥18 year of age at Mayo Clinic Rochester or Mayo Clinic Scottsdale at time of informed consent
4. Have a documented diagnosis of EoE per standard guidelines
5. Have histologically active EoE (defined as a peak eosinophil count >15 eosinophils per high-power field; eos/hpf)
6. Weight ≥40 kg
7. Ability to take injectable or oral medication and be willing to adhere to the study intervention regimen
8. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 12 weeks after the end of dupilumab or budesonide suspension administration. Willingness to complete pregnancy tests during study visits and at end of study.
9. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
10. Subject agrees to maintain a stable diet
11. Subject is willing to receive weekly injections throughout the study
12. Subject is willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Inability to provide informed consent
2. Pregnancy or lactation
3. Contraindication to performing upper endoscopy
4. Known allergic reactions to components of dupilumab or budesonide suspension
5. Non-EoE eosinophilic GI diseases (EGIDs) or hypereosinophilic disorders
6. Prior esophageal surgery, coagulopathy or esophageal varices
7. Known achalasia, crohn's disease, ulcerative colitis, celiac disease
8. Child-Pugh Class C liver disease
9. Failed dupilumab
10. Failed swallowed topical budesonide
11. Erosive esophagitis LA B and above found during EGD
12. Use of prednisone within 2 months prior to study enrollment
13. Treatment with biologic therapies for other disease indications
14. Treatment with medium or high potency topical steroids for skin conditions
15. Autoimmune conditions including lupus, rheumatoid arthritis and psoriatic arthritis
16. Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Esophageal diameter | from enrollment until up to 14 weeks
  the minimum esophageal diameter after 12 weeks of treatment.

SECONDARY OUTCOMES:
Distensibility and diameter change | from baseline to end of treatment at 14 weeks
  Secondary outcomes will include distensibility and change in minimum diameter as measured by endoFLIP topography
EEsAI questionnaire scores | from enrollment to the end of treatment at 12 weeks
  comparison of questionnaires that are scored 0-100 before and after treatment.
Endoscopic refernece score (EREFS) | from enrollment up to end of treatment at 12 weeks
  comparison of EREFs scores on scale of 0-9 at EGDs
Eosinophil counts | from enrollment to the end of treatment at 12 weeks
  number of eosinophils found in biopsy during EGD
Eoe Histologic Scoring system (EoEHSS) | from enrollment to end of treatment at 12 weeks
  An EoEHSS score is given by looking at a biopsy taken during an endoscopy. The score is based on observation of the appearance of the biopsy under a microscope. Score range is 0 to 1
M2 macrophage polarization | from enrollment to end of treatment at 12 weeks
  comparison of myofibroblast differentiation
Lamina propria remodeling | from enrollment to end of treatment at week 12
  characterizing Lamina propria remodeling by second harmonic imaging microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Diana Snyder, M.D., Principal Investigator — Mayo Clinic; Jennifer Horsley-Silva, M.D., Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No